CLINICAL TRIAL: NCT02746848
Title: Evaluation the Effect of Amniotic Membrane Extract Eye Drop (AMEED) on Human Corneal Epithelium Healing (Phase I and II Clinical Trial)
Brief Title: Utilization of Amniotic Membrane Extract Eye Drop (AMEED) on Human Corneal Healing
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Royan Institute (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Royan-Eye-003
Record Dates: First submitted 2016-04-10; First posted 2016-04-21 (Estimated); Last update posted 2016-04-21 (Estimated); Status verified 2016-01

CONDITIONS: Cornea Injury
Keywords: cornea epithelium healing Amniotic Membrane Eye Drop
MeSH Terms: conditions — Corneal Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Patients with cornea injury (Experimental): Patients with cornea injury who received healing Amniotic Membrane Extract Eye Drop.
  Interventions: Biological: Amniotic Membrane Extract Eye Drop

INTERVENTIONS:
Biological: Amniotic Membrane Extract Eye Drop — Amniotic Membrane Extract use as eye drop for patients with corneal injury.

SUMMARY:
For severe ocular surface diseases, such as chemical and thermal injuries, Stevens-Johnson syndrome (SJS), Band Keratopathy, Corneal Dystrophies, Refractive (PRK-LASEK), corneal surgery and others, it is important that short time treatment with minimal side effect should be considered. This study is a prospective clinical trial to use Amniotic Membrane Extract Eye Drop (AMEED) as a natural substance for acceleration of corneal healing

DETAILED DESCRIPTION:
The cornea is the specific anterior part of eye that is essential for normal vision. The corneal surface is comprised of a unique type of non-keratinized epithelial cell. Corneal epithelium contains transient amplifying cells and post mitotic cells. The limbal stem cells (LSC) are located between limbal cornea and conjunctiva which are main source of corneal epithelium healing in eye injuries. For some corneal disease such as chemical and thermal injuries, Corneal Dystrophies and corneal surgery, treatment in short time is important.

AM can modulate corneal epithelium healing by promoting re-epithelialization and migration of limbal stem cell while suppressing stromal inflammation, angiogenesis and scarring. This biological substrate maintain epithelial progenitor cells within the limbal stem cell niche and facilitate ocular surface epithelial renewal. It is well accepted that amniotic membrane Transplantation (AMT) as a temporary patch normally dissolves within 2 weeks. Consequent reapplication of membrane is difficult for the patient.

Other studies have been reported that processed AM as a liquid has comparable effect to AMT in treatment of corneal epithelial healing.

This study is a prospective clinical trial to use Amniotic Membrane Extract Eye Drop (AMEED) as a natural substance for acceleration of corneal healing.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with corneal epithelium injury
2. Without keratoconus
3. Without cornea scar
4. Without any other lesion of cornea

Exclusion Criteria:

1. Lack of timely referral of patients for examinations
2. Simultaneous use of other drugs that cause impairment of the data
3. Previous cornea surgery
4. Dry eye
5. Glaucoma

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2014-06; Primary Completion 2015-05 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
corneal defect size | 12 months
  Evaluation the corneal defect size (millimeter) by microscope after corneal surgery and compare the change of defect size after procedure in compare with base line (before surgery).

SECONDARY OUTCOMES:
Eye Discharge | 1 week
  Evaluation the presence of any abnormal discharge from treated eye after procedure based on side effect questionnaire that fill with patients.
pain | 24 hours
  Evaluation of any presence of pain in treated eye after procedure based on side effect questionnaire that fill with patients.

CONTACTS AND LOCATIONS:
Overall Officials: Hamid Gourabi, PhD, Study Chair — Head of Royan Institute; Marzieh Ebrahimi, PhD, Study Director — Department of Regenerative Biomedicine at Cell Science Research Center, Royan Institute for Stem Cell Biology and Technology, ACECR, Tehran, Iran.; Khosro Jadidi, MD, Study Director — Bina Hospital, Research & Education Center, Tehran, Iran; Fatemeh Doostmohammadi, MD, Principal Investigator — Bina Hospital, Research & Education Center, Tehran, Iran

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://royaninstitute.org